CLINICAL TRIAL: NCT02006849
Title: ACTH Treatment of APOL1- Associated Nephropathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enrollment
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024943
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2016-04

CONDITIONS: Kidney Disease
Keywords: AfricanAmericans; Hypertension; Proteinuria; ApoL1 gene
MeSH Terms: conditions — Kidney Diseases; Hypertension; Proteinuria | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acthar 40 units (Other): Acthar 40 units subcutaneously three times a week for patients with sub-nephrotic proteinuria.
  Interventions: Drug: Acthar
- Acthar 80 units (Other): Acthar 80 units subcutaneously twice a week for patients with nephrotic proteinuria.
  Interventions: Drug: Acthar

INTERVENTIONS:
Drug: Acthar — FDA approved drug being used in this study for sub-nephrotic proteinuria. Given Investigational New Drug (IND) exemption by FDA.
  Other Names: Repository Corticotropin

SUMMARY:
The purpose of this research study is to determine if the study drug H.C. Acthar gel slows the progression of your kidney disease. This drug is a steroid-based medicine with fewer side effects than other steroids used for treatment of kidney diseases similar to APOL1 nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Non-diabetic African-American with two APOL1-risk genotypes
* Age ≥21 years
* BMI < 40 kg/m2
* Hemoglobin A1c <6.5%
* eGFR ≥30 ml/min/1.73m2
* Historical urine protein: creatinine ratio ≥ 1.0 g/g
* Strong clinical suspicion of APOL1-associated nephropathy or history of biopsy proven focal segmental glomerulosclerosis (FSGS) or focal global glomerulosclerosis (FGGS)
* Women of childbearing potential: negative serum pregnancy test at Screening and agreement to follow a medically acceptable form of contraception for the duration of Acthar administration and 4 weeks thereafter

Exclusion Criteria:

* Diagnosis of diabetes mellitus and/or on pharmacologic treatment for diabetes
* Medical condition that could cause secondary FSGS
* History of sensitivity to steroids (psychosis, steroid-induced diabetes)
* Chronic systemic corticosteroid use (Prednisone or equivalent systemic steroid taken for more than 4 consecutive weeks within 6 months prior to screening). Intra-articular, inhaled, and topical steroids are not exclusion criteria.
* Contraindication to Acthar per package insert: scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery (within previous 6 months), history of or the presence of peptic ulcer (within 6 months prior to Screening), adrenal insufficiency or hyperfunction.
* Acute glaucoma diagnosed ≤3 months prior to Screening
* Biopsy proven glomerular disease other than FSGS or FGGS
* Live or live attenuated vaccine received within 1 month prior to screening, or planned administration once enrolled in the study
* Uncontrolled hypertension (HTN) (≥ 180/110 mmHg) and frequent admissions (≥1 admission per 6 months interval) for hypertensive urgency or hypertensive emergency
* Unstable cardiovascular disease: history of congestive heart failure (NYHA Functional Class III-IV); history of dilated cardiomyopathy with ejection fraction < 40%; any of the following events within 3 months of screening: unstable angina, myocardial infarction, coronary artery bypass graft or percutaneous transluminal coronary angioplasty, transient ischemic attack or cerebrovascular accident, unstable arrhythmia
* Uncontrolled volume overload: history of moderate or severe peripheral edema; on loop diuretics ≥ 120 mg daily of furosemide or ≥ 3.0 mg daily of bumetanide or ≥ 150 mg daily of ethacrynic acid or ≥ 60 mg daily of torsemide;
* History of secondary hypertension (i.e., renal artery stenosis, primary aldosteronism or pheochromocytoma)
* Significant comorbidities (e.g., advanced malignancy, advanced liver disease) with a life expectancy of less than 1 year
* Subject is expected to initiate dialysis within 6 months
* Previous treatment on a drug being investigated for the treatment of FSGS
* Known diagnosis of Human Immunodeficiency Virus, Hepatitis B, or Hepatitis C
* Known history of a primary immunodeficiency or an underlying condition such as splenectomy that predisposes the subject to infections
* Systemic hematologic disease (e.g., hematologic malignancy, sickle cell anemia, myelodysplastic syndrome)
* Current malignancy or history of malignancy within 5 years of screening, with the exception of non-melanoma skin cancers and cervical intraepithelial neoplasia
* Treatment for any malignancy (e.g., radiation, chemotherapy, hormone therapy, or biologics) within 5 years of screening, with the exception of locally excised non-melanoma skin cancer or cervical intraepithelial neoplasia
* Pregnant or breast feeding, or might become pregnant during the study or within 4 weeks after the end of treatment
* Female of reproductive potential not willing to use highly effective methods of birth control during treatment and for 4 weeks after the end of treatment
* Currently receiving systemic antibiotics for treatment of an active infection; or history of frequent infections (more than one event per 6 months)
* History of any organ transplant
* Bipolar disorder, or Major Depressive Disorder characterized by severe depression requiring hospitalization, or history of suicidal ideation/attempts
* Currently enrolled in another interventional study, or less than 4 weeks since ending another interventional study(s) or receiving investigational agents(s)
* Subject has a disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with all required study procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in proteinuria with H.C. Acthar gel | End of treatment with H.C. Acthar gel (end of 6 months or 1 year of treatment)
  Complete remission (CR) (UPCR <0.2g/g) or partial remission (PR) (50% drop in UPCR from baseline) of proteinuria at the end of Treatment period in patients with baseline nephrotic proteinuria
Change in proteinuria with H.C. Acthar gel | End of treatment with H.C. Acthar gel (end of 6 months or 1 year of treatment)
  Percent change in proteinuria at the end of Treatment period in patients with baseline sub-nephrotic proteinuria
Change in eGFR with H.C. Acthar gel | End of treatment with H.C. Acthar gel (end of 6 months or 1 year of treatment)
  Percent change in Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) eGFR at the end of Treatment period

SECONDARY OUTCOMES:
Percent change in proteinuria | 1 year and 2 years of study follow-up after treatment completion
  Percent change in proteinuria after 1 year and 2 years of follow-up
Percent change in CKD-EPI eGFR | 1 year and 2 years of study follow-up after treatment completion
  Percent change in CKD-EPI eGFR at 1 and 2 years of study follow-up
Change in CKD-EPI eGFR | 1 year and 2 years of study follow-up after treatment completion
  Change in eGFR over time, based on baseline proteinuria (nephrotic vs. sub-nephrotic), baseline eGFR (eGFR 30-45 vs. eGFR 45-59), and Acthar dose
Duration of remission after H.C. Acthar gel treatment | 1 year and 2 years of study follow-up after treatment completion
  Proportion of patients with baseline nephrotic proteinuria who sustained CR or PR at 1 and 2 years of study follow-up
Changes in kidney fibrosis after H.C. Acthar gel treatment | End of treatment with H.C. Acthar gel (end of 6 months or 1 year of treatment)
  Modifications in kidney histopathology on second post-treatment kidney biopsy (% glomerulosclerosis, % tubulointerstitial fibrosis, restoration of podocyte markers [e.g.,podocin, synaptopodin, Wilms tumor 1]) compared with baseline biopsy
Cholesterol and lipoprotein profile before and after treatment with H.C. Acthar gel | End of treatment with H.C. Acthar gel (end of 6 months or 1 year of treatment)
  Changes in cholesterol and lipoprotein levels compared with baseline profiles

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Murea, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States